CLINICAL TRIAL: NCT07296328
Title: Effects of Psilocybin on Speech Fluency, Struggle, and Brain Activity in People Who Stutter
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-00244
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Stuttering
Keywords: Stuttering; Psilocybin; Stutter
MeSH Terms: conditions — Stuttering | interventions — Psilocybin; Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adult stutterers (Experimental): Participation will occur over an 8-week, 10-session period. Six sessions speech therapy; one preparatory therapy session prior to the drug administration session; one 8-hour drug administration session (25 mg of psilocybin); two follow-up therapy sessions following the drug administration session.
  Interventions: Drug: Psilocybin; Behavioral: Speech therapy

INTERVENTIONS:
Drug: Psilocybin — Participants will receive a single oral high-dose of psilocybin, 25 mg.
Behavioral: Speech therapy — Speech therapy will consist of standard stuttering modification therapy, which includes four phases: Identification, Desensitization, Modification, Stabilization.

SUMMARY:
This Phase 2a clinical trial is an open-label, single-group, within-subjects pilot study designed to evaluate the safety, feasibility, and preliminary efficacy of psilocybin as a therapeutic intervention for adults with developmental stuttering. This pilot study will assess whether further research to explore the potential benefits of psilocybin-assisted therapy for improving clinical outcomes in individuals who stutter, is warranted. The aims of this study include:

* Aim 1: Assess the safety and feasibility of psilocybin as a therapeutic agent for stuttering.
* Aim 2: Evaluate the effects of psilocybin on objective and subjective measures of stuttering severity, struggle, and well-being.
* Aim 3: Explore the therapeutic neural mechanisms of psilocybin in stuttering.

ELIGIBILITY:
Inclusion Criteria:

* Are able to provide voluntary informed consent
* Are able to read, speak, and understand English, as documented during the informed consent process.

  o Non-English-speaking subjects will be excluded because the study is using only validated English-language versions of assessment instruments.
* Are 18 to 50 years old, inclusive, at Screening visit.
* Have diagnosis of mild-moderate to severe stuttering based on either the SSI-4 or OASES; also confirmed stuttering by stuttering specialist.
* Are able and willing to adhere to all study requirements, including attending all study visits and therapy sessions, and completing all assessments.
* Agree to refrain from any non-prescribed psychotropic substance or illicit drug use for at least 72 hours prior to investigational product (IP) administration, and for at least 24 hours before each fMRI assessment visit, with the exceptions of nicotine and caffeine. Regarding nicotine, they must agree not to use nicotine for at least 1 hour before and 6 hours following IP administration, and for at least 1 hour before fMRI scans. Regarding caffeine, they must agree to consume approximately their usual amount of caffeine on the morning of Day 0 (prior to IP administration).
* Agree to refrain from taking all non-prescription medications and supplements (nutritional and herbal) for at least 1 week prior to the IP administration session unless approved by the Investigator.
* Can swallow capsules.
* Subjects who are able to become pregnant must comply with the following conditions:

A. Subjects are considered able to become pregnant unless they

1. Do not have a uterus;
2. Are postmenopausal (has had 12 months of natural amenorrhea with a matching clinical profile [age, history of vasomotor symptoms]) prior to Screening Part 2; or
3. Are surgically sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

B. Subjects who are able to become pregnant must

1. Have a negative pregnancy test at Screening (Reassessed at Day 0 (pre-IP administration);
2. Not be currently breastfeeding;
3. Not intend to become pregnant during participation in this study;
4. Agree to use a highly effective form of contraception from the time of Screening until 7 days after the IP Administration Session. Highly effective forms of contraception include:

   1. Consistent and correct usage of established oral contraception;
   2. Injected or implanted hormonal methods of contraception;
   3. Established intrauterine device or intrauterine system;
   4. Bilateral tubal ligation;
   5. Intercourse with a partner who has undergone effective surgical sterilization, provided that partner is the sole sexual partner of the study subject;
   6. Abstinence from penile/vaginal intercourse, if the Investigator determines that the subject can reliably adhere to the plan, based on evaluation of the participant's preferred and usual lifestyle and social circumstances.
5. Agree not to donate or bank eggs from the time of Screening Part 2 until 7 days after the IP Administration Session.

If able to become pregnant or produce viable sperm (male or female), are willing to use approved contraception for duration of the trial.

Exclusion Criteria:

* Pregnancy or lactation.
* Any medical condition that would preclude safe participation in the study, including the following, as determined by medical history review, physical examination, electrocardiogram (ECG), and clinical laboratory tests:

  * Seizure disorder
  * Significantly impaired liver function, defined as 1) alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN); 2) ALT or AST > 3 × ULN with concomitant total bilirubin > 2.0 × ULN; or 3) ALT or AST ≥ 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia.
  * Cardiovascular disease including coronary artery disease, angina, history of arrhythmia (unless a successful ablation has been performed), heart failure, history of heart valve replacement, and history of cerebrovascular accident or transient ischemic attack.
  * Uncontrolled hypertension with systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg. (Note: participants who otherwise meet all eligibility criteria during the screening visit will have 3 opportunities to produce 1 blood pressure reading ≤ 140/90 mmHg (each reading will be collected at least 15 minutes apart). If blood pressure at Screening is consistently elevated (> 140/90 mmHg across all 3 attempts), participants may be referred to their primary care provider (PCP) for management of hypertension. Participants may continue study participation if the Investigator believes that it is likely that hypertension can be controlled prior to the IP administration session, and the patient is able to provide documentation of adequate control (BP < 140/90 mmHg) prior to the PI administration session.)
  * Resting heart rate > 100 bpm (Note: participants will have an opportunity to return once within the 30-day screening window to make 3 additional attempts at a resting heart rate ≤ 100 bpm.).
  * Serious ECG abnormalities (e.g., evidence of ischemia, myocardial infarction, QT interval corrected for heart rate [QTc] prolongation (QTc > 0.450 seconds), arrhythmia, or conduction abnormalities that increase the risk of arrhythmia.
  * Hyperthyroidism
  * Insulin-dependent diabetes
  * Bradycardia (e.g., heart rate <50 bpm)
  * Orthostatic hypotension
  * Schizotypal and paranoid personality disorders
  * Given potential use of diazepam as an ancillary medication, moderate or greater hepatic impairment (Child-Pugh score ≥ 7) is exclusionary.
  * Any other medical condition which precludes safe participation in the study in the medical opinion of the Investigator. (Note: medical history will be updated on Day 0. Those not meeting the criterion may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator.)
* Have any of the following Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) psychiatric disorders, as determined by the Mini International Neuropsychiatric Interview (MINI) and Psychiatric History at the Screening Visit: (Note: psychiatric history will be re-evaluated on Day 0, but the MINI will not be re-administered on Day 0)

  * Lifetime history of schizophrenia spectrum or other psychotic disorder (including substance or medication-induced psychosis or psychosis due to a co-occurring medical condition).
  * Major depressive disorder (MDD)Post traumatic stress disorder (PTSD)
  * Cluster B personality disorders (antisocial personality disorder, borderline personality disorder, histrionic personality disorder, and narcissistic personality disorder)
  * Bipolar I disorder, Bipolar II disorder, and Cyclothymic disorder
* Have active suicidal ideation with intent, based on Columbia-Suicide Severity Rating Scale (C-SSRS) assessment (severity score > 3) at the Screening visit, confirmed by the Investigator. (Note: this criterion will be reassessed at each visit that occurs prior to Day 0, and on Day 0. Participants will be discharged if actively suicidal, and appropriate follow-up will be arranged.
* Have made a medically significant suicide attempt (i.e., one that had a significant possibility of causing death or permanent harm in the absence of intervention) within the past 12 months, based on Screening C-SSRS assessment and confirmation by the Investigator. (Note: this criterion will be reassessed at each visit that occurs prior to Day 0, and on Day 0. Participants will be discharged if actively suicidal, and appropriate follow-up will be arranged.)
* Have a family history (first degree relatives) of schizophrenia, schizoaffective disorder, or bipolar disorder type 1.
* Have a history of hallucinogen use disorder.
* Have a history of hallucinogen persisting perceptual disorder (HPPD).
* Have any use of classic psychedelics in the past 1 year.
* Have > 25 lifetime uses of classic psychedelics.
* Incarcerated or have pending legal action that could prevent participation in study activities.
* Are unable or unwilling to discontinue taking any protocol-prohibited medications and supplements. (A detailed list of exclusionary medications is found in Section 6.5 of the protocol.) Prohibited medications and supplements must have been stopped for at least 5 elimination half-lives or 14 days, whichever is longer, prior to Day 0 (Note: Psychiatric medications will not be discontinued or changed in order to allow study participation. Concomitant medications will be reassessed on Day 0. Any patient who has started prohibited medications will be discharged from the study.)
* Have a known allergy or hypersensitivity to psilocybin or any of the materials contained in the IP used in the study.
* Have an allergy, hypersensitivity, or other contraindication that would preclude safe treatment of acute hypertension, anxiety, or psychotic symptoms if necessary, during or immediately after the IP Administration Session, using the adjunctive medications used in this pilot study to treat these symptoms (i.e., unable to take captopril and unable to take clonidine; unable to take diazepam; or unable to take olanzapine).
* Have any other medical, psychiatric, or psychosocial disorder, symptom, condition, or situation that is likely to interfere with the establishment of rapport, adherence to study requirements, or safe administration of psilocybin or functional magnetic resonance imaging (fMRI) scanning, based on the judgement of the Investigator. (Note: This criterion will be reassessed on Day 0. Those not meeting the criterion will not be randomized but may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator.)
* Inability to safely complete fMRI sessions (MRI screening form)
* Any history of severe traumatic brain injury (assessed using the Ohio State University Traumatic Brain Injury Identification Method (OSU TBI-ID) modified). (Note: If current (past 12 months) mild/moderate Traumatic Brain Injury (TBI) and Central Sensitization Inventory (CSI) score >/= 12 (for either lifetime month or current month), the PI will determine eligibility.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Stuttering Severity Instrument - 4th Edition (SSI-4) total score | Week 4, Week 12
  The Stuttering Severity Instrument-4th Edition (SSI-4) provides a total score that is compared to age-specific norms to determine severity, with ranges for "Very Mild" to "Very Severe". The SSI-4 calculates individual scores for frequency (2-18), duration (2-18), and physical concomitants (0-20). These individual scores are combined to create a total score, which is then ranked against norms to provide a verbal severity descriptor, such as mild, moderate, severe, or very severe.
Change in frequency subcomponent score of the SSI-4 | Week 4, Week 12
  The Stuttering Severity Instrument-4th Edition (SSI-4) provides a total score that is compared to age-specific norms to determine severity, with ranges for "Very Mild" to "Very Severe". The SSI-4 calculates individual scores for frequency (2-18), duration (2-18), and physical concomitants (0-20). These individual scores are combined to create a total score, which is then ranked against norms to provide a verbal severity descriptor, such as mild, moderate, severe, or very severe.
Change in duration subcomponent score of the SSI-4 | Week 4, Week 12
  The Stuttering Severity Instrument-4th Edition (SSI-4) provides a total score that is compared to age-specific norms to determine severity, with ranges for "Very Mild" to "Very Severe". The SSI-4 calculates individual scores for frequency (2-18), duration (2-18), and physical concomitants (0-20). These individual scores are combined to create a total score, which is then ranked against norms to provide a verbal severity descriptor, such as mild, moderate, severe, or very severe.
Change in physical concomitants subcomponent score of the SSI-4 | Week 4, Week 12
  The Stuttering Severity Instrument-4th Edition (SSI-4) provides a total score that is compared to age-specific norms to determine severity, with ranges for "Very Mild" to "Very Severe". The SSI-4 calculates individual scores for frequency (2-18), duration (2-18), and physical concomitants (0-20). These individual scores are combined to create a total score, which is then ranked against norms to provide a verbal severity descriptor, such as mild, moderate, severe, or very severe.
Change in Overall Assessment of the Speaker's Experience of Stuttering - Adults (OASES-A) score | Week 4, Week 12
  The OASES-A is a tool used by speech-language pathologists to measure the adverse impact of stuttering on an adult's life. It consists of 100 questions rated on a 5-point scale (1-5). The scores from individual questions are added together to create an overall score. The total score is then used to determine the "Impact Rating" on a scale from mild to severe. Higher scores indicate higher levels of negative impact.

SECONDARY OUTCOMES:
Change in self-reported stuttering severity Wright and Ayre Stuttering Self-Rating Profile (WASSP) score | Week 4, Week 12
  The WASSP produces a profile of scores across five subscales. There is a total of 26 items each scored on a seven-point Likert-type scale. A score of '1' represents the least severe/negative perception, while a '7' represents the most severe/negative perception on each scale. Total scores range from 26-182, with higher scores indicating a greater negative impact of stuttering on their life.
Change in the Brief Version of the Unhelpful Thoughts and Beliefs About Stuttering Scales (UTBAS-6) total score | Week 4, Week 12
  The UTBAS-6 is a six-item screening questionnaire for adults who stutter to measure unhelpful thoughts and beliefs associated with speech anxiety. The UTBAS-6 has a subscale score range of 6 to 30 and a total score range of 18 to 90. A higher score indicates more frequent unhelpful thoughts and greater anxiety related to stuttering.
Change in Brief Fear of Negative Evaluation Scale (BFNE-S) total score | Week 4, Week 12
  The BFNE-S consists of 8 items that are rated on a five-point likert scale from 1 (not at all characteristic) to 4 (extremely characteristic). Scores range from 0 to 32. A score of 25 or higher may indicate clinically significant social anxiety.
Change in the Social Interaction Anxiety Scale (SIAS) score | Week 4, Week 12
  The SIAS is a 20-item self-report questionnaire that measures the severity of social anxiety. Each item is rated from 0 (not at all characteristic or true of me) to 4 (extremely characteristic or ture of me). Scores can range from 0 (no social anxiety) to 80 (maximum social anxiety). A score of 36 or higher is often considered clinically significant, suggesting the presence of social anxiety.
Change in Stuttering Anticipation Scale (SAS) score | Week 4, Week 12
  The SAS is a 25-item self-report tool measuring specific action responses (avoidance, physical changes, approach) on a 7-point scale from 1 (Never) to 7 (always). Scores range from 25-175, with higher scores indicating more frequent anticipatory behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bogenschutz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Michael.bogenschutz@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Michael.bogenschutz@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.